CLINICAL TRIAL: NCT06866873
Title: Safety and Feasibility Study of CD19 Chimeric Antigen Receptor (CAR) T Cells in Children with Relapsed or Refractory CD19 Positive Acute Lymphoblastic Leukemia or Lymphoma
Brief Title: CD-19 CAR-T Cell for Pediatric ALL or Lymphoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Children's Hospital (Other)
Responsible Party: Principal Investigator, Cheuk Ka Leung Daniel, Consultant, Hong Kong Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKCH-REC-2021-032
Record Dates: First submitted 2025-03-03; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Lymphoma, B-Cell; Acute Lymphoblastic Leukemia, Pediatric
Keywords: CAR-T cell; Pediatric
MeSH Terms: conditions — Lymphoma, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T cell therapy (Experimental): CAR-T cell infusion intravenously once
  Interventions: Biological: CAR-T

INTERVENTIONS:
Biological: CAR-T — CAR-T cell (CHXCART01) infusion intravenously once at a dose of 0.2-2 million cells/kg recipient body weight

SUMMARY:
This study seeks to examine the efficacy and safety of the administration of autologous T cells that have been modified through the introduction of a chimeric antigen receptor (CAR) targeting the B cell surface antigen CD19 following administration of chemotherapy lymphodepletion regimen in children with relapsed or refractory acute lymphoblastic leukemia (ALL) or lymphoma. The overall goal of this study is to validate the safety profile of administration CD19-CAR T cells and describe the response rate in children with relapsed/refractory ALL or lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have relapsed or refractory ALL or lymphoma treated with at least two lines of therapy. Disease must have either progressed after the last regimen or presented failure to achieve partial or complete remission with the last regimen.
* The patient's disease must be CD19 positive, either by immunohistochemistry or flow cytometry analysis on the last biopsy available.
* Age 1-17 years.
* Performance status: Subjects > 10 years of age: Karnofsky ≥ 50%; Subjects ≤ 10 years of age: Lansky scale ≥ 50%.
* Normal organ function.

  * Total bilirubin ≤ 3 times upper limit of normal
  * AST (SGOT) ≤ 5 times upper limit of normal
  * ALT (SGPT) ≤ 5 times upper limit of normal
  * Serum Creatinine ≤ 2 times upper limit of normal
  * Subjects must have the following hematologic function parameters: Hemoglobin (Hb) level > 8 g/dL; Absolute Lymphocyte Count > 0.1x10^9/L; Platelet > 50x10^9/L
* Prior therapy wash-out. At least 2 weeks or 5 half lives, whichever is shorter, must have elapsed since any prior systemic therapy at the time the subject is planned for leukapheresis.
* Subjects' parent or legal guardian must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Autologous transplant within 6 weeks of planned CAR T cell infusion.
* Recipient of CAR-T cell therapy outside of this protocol.
* Active central nervous system (CNS) or meningeal involvement by tumor.
* History of additional active malignancy other than non-melanoma skin cancer, carcinoma in situ (e.g. cervix, bladder, breast).
* Active human immunodeficiency virus (HIV) infection.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary abnormalities or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women.
* Evidence of myelodysplasia or cytogenetic abnormality indicative of myelodysplasia on any bone marrow biopsy prior to initiation of therapy.
* Serologic status reflecting active hepatitis B or C infection.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2037-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CRR) for ALL and Overall response rate (ORR) for lymphoma | 1 month for subjects with ALL, and 3 months for subjects with lymphoma
  Complete response for ALL was defined as leukemic cells <5% in bone marrow. Overall response for lymphoma was defined as complete response plus partial response defined by Lugano criteria.
Incidence and severity of adverse events | through study completion, an average of 6 months
  Severity of adverse events are graded according to CTCAEv5.0.

SECONDARY OUTCOMES:
Frequency of minimal residual disease for ALL | 1 month
  Measurable residual disease in bone marrow by flow cytometry or PCR methods.
Overall survival | 1 year
  survival as estimated by Kaplan-Meier method. Death from any cause is considered as event for analysis.
Event-free survival | 1 year
  Event-free survival as estimated by Kaplan-Meier method. Events are death from any cause, or relapse or progression of underlying disease.
Proportion of products successfully manufactured | at the time of CAR-T cell infusion
  Success defined as meeting product release criteria with at least 0.2 million cells/kg recipient body weight

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Lee, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Hong Kong Children's Hospital, Hong Kong, Hong Kong